CLINICAL TRIAL: NCT03858751
Title: Pharmacological Activation of Hypoglossal Motor Nucleus for Obstructive Sleep Apnea Aim 2
Brief Title: Pharmacological Activation of HMN for OSA Aim 2
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Scott Aaron Sands, Principal investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018p001201aim2
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo capsule before bedtime
  Interventions: Drug: Placebo oral capsule
- LTM1201AZ (Experimental): LTM1201AZ capsule before bedtime
  Interventions: Drug: LTM1201AZ
- LTM1201AT (Experimental): LTM1201AT capsule before bedtime
  Interventions: Drug: LTM1201AT
- LTM1201AG (Experimental): LTM1201AG capsule before bedtime
  Interventions: Drug: LTM1201AG
- LTM1201AD (Experimental): LTM1201AD capsule before bedtime
  Interventions: Drug: LTM1201AD

INTERVENTIONS:
Drug: Placebo oral capsule — Placebo capsule before bedtime
  Arms: Placebo
Drug: LTM1201AZ — LTM1201AZ oral capsule before sleep
  Arms: LTM1201AZ
Drug: LTM1201AT — LTM1201AT oral capsule before sleep
  Arms: LTM1201AT
Drug: LTM1201AG — LTM1201AG oral capsule before sleep
  Arms: LTM1201AG
Drug: LTM1201AD — LTM1201AD oral capsule before sleep
  Arms: LTM1201AD

SUMMARY:
Obstructive sleep apnea (OSA) is common and has major health implications but treatment options are limited. OSA patients show a marked reduction in upper airway (UA) dilator muscle activity at sleep onset and this phenomenon leads to increased collapsibility of UA compared to normal subjects. In this protocol the investigators will test the effect of LTM1201AZ, LTM1201AT, LTM1201AD, LTM1201AG administered before sleep on OSA phenotype traits and OSA severity during sleep.

ELIGIBILITY:
Inclusion Criteria:

* AHI > 10 events/h during NREM supine sleep

Exclusion Criteria:

* Any medical condition other than well controlled hypertension and mild diabetes.
* Any medication known to influence breathing, sleep/arousal, or muscle physiology.
* Claustrophobia.
* Inability to sleep supine.
* Allergy to any of the medications tested in the protocol.
* History of kidney stones, hypercalcemia, primary hyperparathyroidism, sarcoidosis, hypervitaminosis D.
* Individuals with underlying cardiac disease, such as arrhythmias.
* Individuals taking psychiatric medications, such as an MAO-I, SSRI or SNRI, or any of the studied medications for medical care.
* For women: Pregnancy.
* Pulmonary hypertension
* Severe OSA with a mean SaO2 lower than 88%

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Apnea hypopnea Index (AHI, average number of events for every hour of sleep) | 3 nights (treatment duration)
  Based on previous studies the investigators anticipate that active comparators will reduce AHI more effectively in subjects with moderate sleep apnea and low-to-moderate collapsibility (Vpassive >50% of eupneic values). Higher AHI indicates more severe OSA, usually ranging between 10 to 110 events/hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No